CLINICAL TRIAL: NCT01648647
Title: GE DHM-AN-OR-2012/01
Brief Title: Copeptin in Aortic Valve Replacement
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: GE DHM-AN-OR-2012/01
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Copeptin in Patients Undergoing Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Copeptin is accepted as a marker of stress. We want to evaluate the preoperative and early postoperative copeptin leavens in patients undergoing different aortic valve procedures

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical aortic valve replacment
* Patients undergoing transcatheter aortic valve replacment

Exclusion Criteria:

* denial by patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgical or transcatheter aortic valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-05

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum München des Freistaates Bayern, Technische Universität München, Munich, Bavaria, Germany